CLINICAL TRIAL: NCT00452049
Title: Observational Study to Evaluate the Effect of Parathyroidectomy on Renal Function, Endothelial Function and Blood Pressure
Brief Title: The Effect of Parathyroidectomy on Renal Function, Endothelial Function, and Blood Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Evenepoel Pieter, MD, PhD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: ML3052
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Hyperparathyroidism; Hypertension
Keywords: parathyroidectomy; arterial stiffness; renal function
MeSH Terms: conditions — Hyperparathyroidism; Hypertension | interventions — Parathyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: parathyroidectomy — parathyroidectomy

SUMMARY:
Secondary hyperparathyroidism (HPT) is a known complication of chronic renal failure. Elevated concentrations of parathyroid hormone (PTH) play a role not only in the pathogenesis of renal bone disease, but also in the development of cardiovascular risk factors such as disturbed lipid metabolism, glucose intolerance, and hypertension. HPT is also known to play an important role in the development of structural abnormalities of both large arteries and the heart (left ventricular hypertrophy, interstitial fibrosis). In the last couple of years there has been increasing evidence from animal studies that the endothelium is a target organ of PTH.

Hypothesis: PTH has clinically relevant effects on renal hemodynamics, renal function and endothelial function.

Aims:

1. To evaluate the effect of parathyroidectomy (PTX) on renal hemodynamics in stable renal transplant recipients
2. To evaluate the effect of PTX on endothelial function in stable renal transplant recipients/chronic kidney disease (CKD) stage 5 patients
3. To evaluate the effect of PTX on blood pressure in stable renal transplant recipients/CKD stage 5 patients

ELIGIBILITY:
Inclusion Criteria:

1. Stable renal transplant recipients/CKD stage 5D patients.
2. Age between 18 years and 85 years.
3. Signed informed consent.
4. PTX scheduled because of severe hyperparathyroidism (day 0)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Evenepoel, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hopsital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Evenepoel P, Claes K, Viaene L, Bammens B, Meijers B, Naesens M, Sprangers B, Kuypers D. Decreased Circulating Sclerostin Levels in Renal Transplant Recipients With Persistent Hyperparathyroidism. Transplantation. 2016 Oct;100(10):2188-93. doi: 10.1097/TP.0000000000001311. PMID 27379556